CLINICAL TRIAL: NCT03755739
Title: A Phase II/III Trial of Comparison of Benefit of Administration of Checkpoint Inhibitors Plus Chemodrug Via Artery or Fine Needle to Tumor Versus Vein for Immunotherapy of Advanced Solid Tumors
Brief Title: Trans-Artery/Intra-Tumor Infusion of Checkpoint Inhibitors Plus Chemodrug for Immunotherapy of Advanced Solid Tumors
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZZITICI-004
Record Dates: First submitted 2018-11-03; First posted 2018-11-28 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Hepatocarcinoma; Lung Cancer; Melanoma; Renal Cancer; Head and Neck Cancer; Pancreas Cancer; Ovarian Cancer; Colo-rectal Cancer; Cervical Cancer; Breast Cancer
Keywords: Solid cancers; Check-point inhibitors; Interventional Radiology; Trans-artery infusion; Intra-tumor injection
MeSH Terms: conditions — Carcinoma, Hepatocellular; Lung Neoplasms; Melanoma; Kidney Neoplasms; Head and Neck Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Colonic Neoplasms; Uterine Cervical Neoplasms; Breast Neoplasms | interventions — cyclopropapyrroloindole; pembrolizumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pembrolizumab via localized infusion (Experimental): This group dividied into two subgroups:
  1. Checkpoint inhibitor (CPI) such as Pembrolizumab ± Ipilimumab is administrated with a dose of 1-2mg/kg via sustained (10min) micro-pump infusion via artery, plus chemotherapy, every 3 weeks.
  2. Checkpoint inhibitor (CPI) such as Pembrolizumab ± Ipilimumab is administrated with a total dose of 150mg via intra-tumor fine needle injection in 5 min, plus doxorubicin, every 3 weeks.
  Interventions: Drug: Checkpoint inhibitor (CPI) such as Pembrolizumab plus chemotherapy
- Checkpoint inhibitor (CPI) Pembrolizumab plus chemotherapy via vein infusion (Active Comparator): Checkpoint inhibitor (CPI) such as Pembrolizumab is administrated with a total dose of 2mg/kg via vein infusion (30 min), plus chemotherpy every 3 weeks.
  Interventions: Drug: Checkpoint inhibitor (CPI) such as Pembrolizumab plus chemotherapy

INTERVENTIONS:
Drug: Checkpoint inhibitor (CPI) such as Pembrolizumab plus chemotherapy — vein, artery, or intra-tumor infusion of checkpoint inhibitor (CPI) such as Pembrolizumab and/or Ipilimumab, plus chemotherapy to destroy cancer cells and release tumor antigen for improving CPI therapeutic efficacy.
  Other Names: Checkpoint inhibitor (CPI) such as Keytruda plus chemotherapy

SUMMARY:
This trial was designed to investigate the safety, response rates and survival outcomes of patients with advanced solid tumors by trans-artery/intra-tumor infusion of PD1/PDL1 antibody and/or CTLA4 antibody ipilimumab plus chemotherapeutic drug and to compare their differences.

DETAILED DESCRIPTION:
Malignant solid tumors including lung and liver cancers are the most common malignancy worldwide, and their mortality rates are very high. China has a huge population base, with about 4,000,000 new cases each year. More than 60% of the solid tumors in China are diagnosed at mid-to-late stage and have lost the chance of surgery. Recently a lot of therapeutic strategies have been developed and applied to clinic including targeted therapy and immunotherapy, but the overall efficiency is still low. It is difficult to be widely used in patients with advanced solid cancers, and more alternative therapies are urgently needed.

Antibodies against PD1, PDL1 and CTLA4 are representative drugs for the check-points inhibitory agents, and their clinical indications have been approved in various types of tumors, including advanced melanoma, non-small cell lung cancer, renal cell carcinoma, and classical Hodgkin's lymphoma and late recurrent head and neck squamous cell carcinoma patients, et al. Those drugs are regularly systemically administrated by vein infusion, however, local delivery of those drugs via interventional radiology technique including trans-artery or intra-tumor injection may increase the local drug concentration in the tumor, improve the efficacy, and reduce systemic adverse reactions, through so called "first pass effect" of drug on target organs. To the investigator's knowledge, no studies have been developed on the efficacy and survival benefit of localized delivery of checkpoint inhibitors for treatment of cancer patients. This phase II-III clinical trial was designed to compare the effects of Pembrolizumab, Tecentriq, et al and/or ipilimumab plus chemotherapeutic drug such as doxorubicin on the survival benefit of patients with advanced solid cancers, including ORR, DCR, median survival time, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Cytohistological confirmation is required for diagnosis of cancer.
2. Signed informed consent before recruiting.
3. Age above 18 years with estimated survival over 3 months.
4. Child-Pugh class A or B/Child score > 7; ECOG score < 2
5. Tolerable coagulation function or reversible coagulation disorders
6. Laboratory examination test within 7 days prior to procedure: WBC≥3.0×10E9/L; Hb≥90g/L； PLT ≥50×10E9/L；INR < 2.3 or PT < 6 seconds above control；Cr ≤ 145.5 umul/L；Albumin > 28 g/L；Total bilirubin < 51 μmol/L
7. At least one tumor lesion meeting measurable disease criteria as determined by RECIST v1.1.
8. Birth control.
9. Willing and able to comply with scheduled visits, treatment plan and laboratory tests.

Exclusion Criteria:

1. Patients participated in clinical trials of equipment or drugs (signed informed consent) within 4 weeks;
2. Patients accompany by ascites, hepatic encephalopathy and esophageal and gastric varices bleeding;
3. Any serious accompanying disease, which is expected to have an unknown, impact on the prognosis, include heart disease, inadequately controlled diabetes and psychiatric disorders;
4. Patients accompanied with other tumors or past medical history of malignancy;
5. Pregnant or lactating patients, all patients participating in this trial must adopt appropriate birth control measures during treatment;
6. Patients have poor compliance.

   Any contraindications for hepatic arterial infusion procedure:

   A.Impaired clotting test (platelet count < 60000/mm3, prothrombin activity < 50%).

   B.Renal failure / insufficiency requiring hemo-or peritoneal dialysis. C.Known severe atheromatosis. D.Known uncontrolled blood hypertension (> 160/100 mm/Hg).
7. Allergic to contrast agent;
8. Any agents which could affect the absorption or pharmacokinetics of the study drugs
9. Other conditions that investigator decides not suitable for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2033-11-01 (Estimated); Study Completion 2036-11-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Overall survival (OS) will be defined as the elapsed time from the enrollment to death from any cause. For surviving patients, follow-up will be censored at the date of last contact (or last date known to be alive). Follow-up for OS will occur every 12 weeks (±1 month) until death or withdrawal of consent from the study.
Complete response (CR) rate before or at Month 6 | 4
  Percentage of patients achieving complete response (CR) before or at Month 6

SECONDARY OUTCOMES:
Progression-free survival | 5 years
  Progression-free survival (PFS) will be defined as the elapsed time from the first date of study treatment until documented disease progression (as per mRECIST) or death from any cause, whichever is earlier. For patients who remain alive without progression, follow-up time will be censored at the date of last disease assessment.
Duration of remission (DOR) | 5 years
  DOR will be defined as the duration of the cancer remission
Disease control rate | 5 years
  Disease control rate will be defined as objective response rate + steady disease rate.
Cause of death (COD) when appropriate | 5
  Cause of death (COD) when appropriate

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD,PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tan H, Shah NUH, He B, Liu T, Li T, Liu M, Gu Y, Zhi C, Ou Y, Huang J, Li M, Zuo S, Chen D, Qin R, Yang H, Li X, Lian H, Wu Q, Leidner R, Chen R, Yang A, Yang L, Zhang Z. Intratumoral delivery of PD-1/PD-L1 and CTLA-4 inhibitors for recurrent/refractory solid tumors: a proof-of-concept treatment strategy. Front Immunol. 2025 Dec 12;16:1669924. doi: 10.3389/fimmu.2025.1669924. eCollection 2025. PMID 41459523